CLINICAL TRIAL: NCT00176800
Title: Pre-Operative Chemoradiation Followed by Post-Operative Tetrathiomolybdate (TM) in Patients With Loco-Regional Esophageal Carcinoma (UMCC 2001-007)
Brief Title: Chemoradiation and Tetrathiomolybdate (TM) in Patients With Esophageal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2001-007; HUM 49005 Legacy 2001-0623 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Esophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — tetrathiomolybdate; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Paclitaxel is administered intravenously over 1 hour on Days 1, 8, 15, and 22. Cisplatin will then be administered intravenously over 1 hour on Days 1 and 22. Radiation treatments will be given twice/day, on Days 1-5, 8-12 and 15-19. The subject's esophagus will be surgically removed on approximately Day #50. Approximately 4-6 weeks after surgery, the subject will start taking Tetrathiomolybdate, for 2 years or until treatment is no longer working to control your cancer. The subject will have blood drawn weekly while he/she is receiving chemotherapy and radiation prior to their surgery. 4-6 weeks after their surgery (when the subject starts taking Tetrathiomolybdate), a blood test will be performed every other week for 2 times, and monthly thereafter. When the level of copper has been lowered sufficiently an additional blood test and a baseline chest x-ray will be obtained. Additional blood will be drawn and tested every 6 months for the first 2 years.
  Interventions: Drug: Tetrathiomolybdate (TM); Procedure: Radiation; Procedure: Surgery

INTERVENTIONS:
Drug: Tetrathiomolybdate (TM) — Tetrathiomolybdate: 20mg p.o. per day with largest meal. This will be started 4-6 weeks post-op, and continued x 2 years or until progression of disease is documented.
Procedure: Radiation — Radiation treatments will be administered twice per day with each dose separated by more than 6 hours, on Days 1-5, 8-12 and 15-19.
Procedure: Surgery — The persons's esophagus will be surgically removed (esophagectomy) on approximately Day #50.

SUMMARY:
Surgery has been the standard of care for esophageal cancer for many years, with limited success. At present, several studies are underway nationwide which utilize chemotherapy combined with radiation therapy prior to the usual surgical regimen. Although this treatment offers some possibility for improvement of patients with esophageal cancer, there remains a significant need for development of new drugs that can substantially impact survival

Investigators at the University of Michigan have been evaluating inhibitors of tumor blood vessel growth (angiogenesis). Specifically, they are evaluating the role of copper in angiogenesis. Copper has been shown to be both a requirement and a potent stimulus for angiogenesis.

Previous studies have shown Tetrathiomolybdate (TM) to rapidly lower copper levels in the blood. The physicians at the University of Michigan are studying whether the addition of TM to the chemoradiation and surgery may increase survival for patients with esophageal cancer.

DETAILED DESCRIPTION:
The pre-study evaluations include a medical history, physical examination, blood laboratory evaluations, and scans to evaluate disease. A CT scan will be performed to measure the size of the subject's tumor(s). The treatment phase of the study includes: 1. Administration of Paclitaxel as an intravenous infusion over 1 hour on Days #1, 8, 15, and 22. 2. Cisplatin will be given as an intravenous infusion after Paclitaxel over 1 hour on Days #1 and 22. 3. Radiation treatments twice per day with each dose separated by more than 6 hours, on Days 1-5, 8-12 and 15-19.

The subject's esophagus will be surgically removed (esophagectomy) on approximately Day #50.

Approximately four to six weeks after surgery, the subject will start taking Tetrathiomolybdate, one pill a day by mouth, for two years or until treatment is no longer working to control your cancer. The dose may need to be increased by 1 pill every 2 weeks, depending on the results of blood tests that are given on a routine basis to help guide the dosing.

Dietary Restrictions: Subjects may not eat shell fish or liver (organ meat) while on study due to high copper content.

Blood draws (approximately 1-2 tablespoons) will be taken weekly while the subject is undergoing chemotherapy and radiation prior to surgery. Prior to your surgery a CT scan will also be administered. Four to six weeks after surgery (when the subject is starting to take Tetrathiomolybdate), a blood test (approximately 1 teaspoon) will be performed every other week for 2 times, and monthly thereafter. This blood test will check for the amount of copper in the subject's blood. When the level of copper has been lowered sufficiently (which will be determined by your physician) an additional blood test and a baseline chest x-ray will be obtained.

Additional blood will be drawn (approximately 1-2 tablespoons) and tested every 6 months for the first 2 years.

There are circumstances under which treatment may be discontinued whether the subject agrees or not. These circumstances include: the subject's tumor gets worse despite the treatment; side effects of the treatment are too dangerous for the subject; new information about the drug becomes available and this information suggests the drug will be ineffective or unsafe for the subject.

ELIGIBILITY:
Eligibility Requirements

1. Histologically confirmed adenocarcinoma or squamous cell carcinoma of the esophagus or gastroesophageal junction
2. No prior treatment for the esophageal cancer allowed.
3. No prior thoracic or upper abdominal radiation.
4. Disease should be limited to the esophagus and regional lymph nodes. Regional lymph nodes are described in Section 4.0. However, celiac node enlargement will be acceptable for tumors of the distal esophagus, because they will be included in the radiation field.
5. Disease must be able to be encompassed in a single radiation field.
6. No medical contraindication to surgery
7. All treatment is to be administered at the University of Michigan Medical Center.
8. Karnofsky Performance Status (scoring system used to quantify general well-being and activities of daily life; scores range from 0 to 100% where 100% represents perfect health and 0 represents death) > 70 %.
9. Age range: 18 - 75 years old.
10. Adequate baseline hematopoetic function:

    Platelet count equal to or greater than 100,000/mm3 Absolute granulocyte count equal to or greater than 1500/mm3 Hematocrit equal to or greater than 29% (patients may be transfused to this level)
11. Adequate baseline organ function :

    Creatinine clearance >/= 60 mls/min Bilirubin equal to or less than 1.5 x upper limits of normal AST (aspartate aminotransferase)/ALT (alanine aminotransferase) equal to or less than 2.5 x upper limits of normal
12. Patients with any complaint of hearing loss should be evaluated with an audiogram. The average pure tone average hearing loss from 500-2000Hz should not exceed 30 dB. If it does, the patient should be warned that further hearing loss may be very noticeable and permanent.
13. Prior malignancy is acceptable if the patient is considered to be cured. In most cases this will mean a 5-year disease-free period. Contact the Principal Investigator for any specific question regarding this requirement.
14. Patients with active infection, serious inter-current medical conditions are ineligible, according to the judgment of the investigators.
15. Pregnant or lactating females are not eligible. Women of childbearing Potential must be using contraception throughout the entire period of treatment.
16. Ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2001-11; Primary Completion 2006-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Urba, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemoradiation and Tetrathiomolybdate (TM): Paclitaxel is administered intravenously over 1 hour on Days 1, 8, 15, and 22. Cisplatin will then be administered intravenously over 1 hour on Days 1 and 22. Tetrathiomolybdate (TM): Tetrathiomolybdate: 20mg p.o. per day with largest meal. This will be started 4-6 weeks post-op, and continued x 2 years or until progression of disease is documented.
  Radiation: Radiation treatments will be administered twice per day with each dose separated by more than 6 hours, on Days 1-5, 8-12 and 15-19.
  Surgery: The persons's esophagus will be surgically removed (esophagectomy) on approximately Day #50.
Period: Overall Study
Arm/Group | Chemoradiation and Tetrathiomolybdate (TM)
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemoradiation and Tetrathiomolybdate (TM)
Number analyzed (Participants) | 69
Age, Continuous [Median (Full Range); unit: years] | 60 [42 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Median Recurrence Free Survival Time
Description: To measure the time recurrence in patients with esophageal cancer treated with preoperative chemoradiation, surgery, and post-operative tetrathiomolybdate.
Time Frame: 8 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemoradiation and Tetrathiomolybdate (TM)
Number analyzed (Participants) | 69
months | 23.1 [12.7 to 60.1]

2. Secondary Outcome: Median Overall Survival Time
Description: To measure the survival time in patients treated with preoperative chemoradiation, surgery, and post-operative tetrathiomolybdate.
Time Frame: 8 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemoradiation and Tetrathiomolybdate (TM)
Number analyzed (Participants) | 69
months | 31.5 [17.1 to 62.4]

3. Secondary Outcome: Percentage of Patients That Require Dose Modification Due to Toxicity
Time Frame: 8 years
Measure: Number; unit: percentage of patients
Arm/Group | Chemoradiation and Tetrathiomolybdate (TM)
Number analyzed (Participants) | 69
percentage of patients
  Leukopenia | 22
  Vomiting | 6

ADVERSE EVENTS:
Arm/Group | Chemoradiation and Tetrathiomolybdate (TM)
Serious Adverse Events (participants affected / at risk) | 28/69
Other Adverse Events (participants affected / at risk) | 67/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation and Tetrathiomolybdate (TM) (N=69)
Anorexia (General disorders) | 2
Bilirubin (Investigations) | 1
Cardiac-ischemia/infarction (Cardiac disorders) | 1
Cardiovascular/Arrhythmia-Other (Cardiac disorders) | 1
Catheter-related infection (Infections and infestations) | 1
Chest pain (non-cardiac and non-pleuritic) (Musculoskeletal and connective tissue disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 1
Diarrhea (no colostomy) (Gastrointestinal disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Gastrointestinal-Other (Gastrointestinal disorders) | 2
Hypokalemia (Investigations) | 1
Hypotension (Cardiac disorders) | 1
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 1
Infection without neutropenia (Infections and infestations) | 2
Melena/GI bleeding (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Operative injury of vein/artery (Injury, poisoning and procedural complications) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 1
Supraventricular arrhythmias (Cardiac disorders) | 1
Thrombosis/embolism (Vascular disorders) | 1
Thrombotic microangiopathy (Vascular disorders) | 2
Wound-non-infectious (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation and Tetrathiomolybdate (TM) (N=69)
Anemia (Blood and lymphatic system disorders) | 31
Leukopenia (Blood and lymphatic system disorders) | 54
Neutopenia (Blood and lymphatic system disorders) | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Nausea (Gastrointestinal disorders) | 30
Vomiting (Gastrointestinal disorders) | 22
Diarrhea (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes